CLINICAL TRIAL: NCT00628498
Title: Defibrotide for Patients With Hepatic Veno-occlusive Disease: A Treatment IND Study
Acronym: Treatment IND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2006-05
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Results first posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Hepatic Veno-Occlusive Disease
Keywords: VOD
MeSH Terms: conditions — Hepatic Veno-Occlusive Disease | interventions — defibrotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Defibrotide (Experimental): Defibrotide 25 mg/kg day given in 4 divided doses approximately every 6 hours
  Interventions: Drug: Defibrotide

INTERVENTIONS:
Drug: Defibrotide — Defibrotide is a single-stranded polydeoxyribonucleotide derived from porcine intestinal mucosa by controlled depolymerisation. Defibrotide has a complex mechanism of action with antithrombotic, anti-ischemic, anti-inflammatory, anti-adhesive and thrombolytic properties but no significant systemic anti-coagulant effects.
  Defibrotide is dose intravenously as a 2-hour infusion every 6 hours at a dose of 25 mg/kg/day. Recommended duration of therapy is 21 days.
Drug: Defibrotide

SUMMARY:
Single arm, open-label study to provide Defibrotide to patients diagnosed with VOD. Defibrotide is no longer available though the Emergency Use IND mechanism (also known as compassionate use, or single patient named use). This protocol is the only mechanism by which Defibrotide can be made available to patients in the U.S.

ELIGIBILITY:
Inclusion Criteria:

Entry criteria include the following:

1. Clinical diagnosis of VOD, made by Baltimore Criteria, Modified Seattle Criteria, or biopsy proven:

   1.1 Baltimore Criteria- Bilirubin ≥2 mg/dL and at least 2 of the following clinical findings:
   * Ascites (radiographic or physical exam)
   * Weight gain of ≥5% compared to the day of conditioning-- if this value is not available, the weight on the date of admission to the SCT unit may be used)
   * Hepatomegaly; increased over baseline.

   1.2 Modified Seattle Criteria: At least two of the following
   * Bilirubin ≥2 mg/dL
   * Ascites (radiographic or physical exam) and/or weight gain ≥5% above baseline weight (defined as weight on the first day of conditioning- if this value is not available, the weight on the date of admission to the SCT unit may be used)
   * hepatomegaly increased over baseline

   1.3 Patients that do not meet the Baltimore Criteria or Modified Seattle Criteria and have biopsy proven VOD are eligible.
2. Patient must also provide written informed consent.

Exclusion Criteria:

* Use of any medication which increases the risk of hemorrhage is disallowed. Use of heparin or other anticoagulants is disallowed within 12 hours unless being used for routine central venous line management, fibrinolytic instillation for central venous line occlusion, intermittent dialysis or ultrafiltration of CVVH.
* Clinically significant uncontrolled acute bleeding, defined as hemorrhage requiring > 15 cc/kg of packed red blood cells (e.g., a pediatric patient weighing 20 kg and requiring > 300cc of packed red blood cells/24 hours, or an adult patient weighing 70 kg and requiring >3 units of packed red blood cells/24 hours) to replace blood loss, OR bleeding from a site which in the Investigator's opinion constitutes a potential life-threatening source (e.g. pulmonary hemorrhage or CNS bleeding), irrespective of amount of blood loss, at any point from the date of SCT through the date of severe VOD diagnosis.
* Hemodynamic instability as defined by a requirement for multiple pressors, or inability to maintain mean arterial pressure (for children: to maintain mean arterial pressure within 1 standard deviation of age-adjusted levels) with single pressor support.
* Woman who are pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1206 (Actual)
Dates: Start 2007-12; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Tappe, M.D., Study Chair — Jazz Pharmaceuticals; Paul Richardson, M.D., Principal Investigator — Dana-Farber Cancer Institute
Locations (125):
- United States (125):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Mayo Clinic Cancer Center, Phoenix, Arizona
  - Arizona Oncology, Scottsdale, Arizona
  - University Medical Center, Tucson, Arizona
  - University of Arkansas for Medical Services, Little Rock, Arkansas
  - City of Hope Medical Center, Duarte, California
  - The University of California, San Diego, La Jolla, California
  - Loma Linda University, Loma Linda, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital & Research Center Oakland, Oakland, California
  - Children's Hospital of Orange County (CHOC), Orange, California
  - Sutter Institute for Medical Research, Sacramento, California
  - University of California Davis Health System, Sacramento, California
  - Rady's Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - US Oncology - Denver, Denver, Colorado
  - Yale - New Haven Hospital, New Haven, Connecticut
  - Nemours-Al duPont Hospital for Children, Wilmington, Delaware
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - UF Health Shands Hospital, Gainesville, Florida
  - Jackson Memorial- University of Miami Health System- Pediatrics, Miami, Florida
  - Nicklaus Children's Hospital (Miami Children's Hospital), Miami, Florida
  - Florida Hospital, Orlando, Florida
  - All Children's Hospital Specialty Physicians, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Childrens Healthcare of Atlanta, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Kapi'olani Medical Center for Women and Children, Honolulu, Hawaii
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwest Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Pediatric Hematology/Oncology MC4060 - University of Chicago, Chicago, Illinois
  - Cardinal Bernardin Cancer-Loyola University Medical Center, Maywood, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Indiana Blood and Marrow Transplantation Clinical Lab LLC/St. Francis Hospital, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Pediatric Blood and Cancer Disorders Clinic, Louisville, Kentucky
  - University of Louisville Research Foundation, Louisville, Kentucky
  - Tulane University Hospital & Clinic (Tuhc) - Tulane Cancer Center Comprehensive Clinic (Tcccc), New Orleans, Louisiana
  - Children's Hospital, New Orleans, Louisiana
  - University of Maryland - Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - National Institutes of Health, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital DFCI/CHB-Pediatrics, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Wayne State University/Children's Hospital of Michigan, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Helen DeVos Children's Hospital - Spectrum Health, Grand Rapids, Michigan
  - Children's Hospitals and Clinics of Minnesota and Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital and Clinics - Infectious Diseases, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center/St. Louis University Department of Pediatrics, St Louis, Missouri
  - Washington University/St. Louis Children's Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center - Joseph M. Sanzari Childrens Hospital, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Presbyterian Hospital, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Steven and Alexandra Cohen Children's Medical Center, New Hyde Park, New York
  - New York University School of Medicine, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Mount Sinai Hospital - BMT Program, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Morgan Stanley Children's Hospital - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York
  - University of Rochester Medical Center, Strong Memorial Hospital, Rochester, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Levine Children's Hospital, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Children's Hospital Medical, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Jewish Hospital, Cincinnati, Ohio
  - Case Western Reserve University (Cwru) - University Hospitals of Cleveland (Uhc), Cleveland, Ohio
  - Robert J Tomsich Pathology & Laboratory Medicine Institute, Cleveland, Ohio
  - Nationwide Children's Hospital - Ohio State University College of Medicine (OSUCOM), Columbus, Ohio
  - The Ohio State University, James Cancer Hospital, Columbus, Ohio
  - The University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Doernbecher Children's Hospital - Oregon Health and Science University, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - West Penn Allegheny Health System, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Methodist University Hospital, Memphis, Tennessee
  - St. Jude Children's Research Hospital - Department of Bone Marrow Transplantation and Cellular Therapy, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Children's Medical Center of Dallas, Dallas, Texas
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - Cook Children's Health Care Hospital, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - The University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Methodist Healthcare System of San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Children's Hospital of the King's Daughter, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center/Seattle Children Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Babb Randolph Cancer Center - West Virginia University Hospital, Morgantown, West Virginia
  - University of Wisconsin, American Family Children's Hospital, Medical School, Madison, Wisconsin
  - Medical College of Wisconsin/ Children's Hospitalof Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Result] Richardson PG, Murakami C, Jin Z, Warren D, Momtaz P, Hoppensteadt D, Elias AD, Antin JH, Soiffer R, Spitzer T, Avigan D, Bearman SI, Martin PL, Kurtzberg J, Vredenburgh J, Chen AR, Arai S, Vogelsang G, McDonald GB, Guinan EC. Multi-institutional use of defibrotide in 88 patients after stem cell transplantation with severe veno-occlusive disease and multisystem organ failure: response without significant toxicity in a high-risk population and factors predictive of outcome. Blood. 2002 Dec 15;100(13):4337-43. doi: 10.1182/blood-2002-04-1216. Epub 2002 Aug 1. PMID 12393437
- [Derived] Richardson PG, Smith AR, Kernan NA, Lehmann L, Ryan RJ, Grupp SA. Analysis of Time to Complete Response after Defibrotide Initiation in Patients with Hepatic Veno-Occlusive Disease/Sinusoidal Obstruction Syndrome after Hematopoietic Cell Transplantation. Transplant Cell Ther. 2021 Jan;27(1):88.e1-88.e6. doi: 10.1016/j.bbmt.2020.09.008. Epub 2020 Sep 17. PMID 32950693
- [Derived] Kernan NA, Grupp S, Smith AR, Arai S, Triplett B, Antin JH, Lehmann L, Shore T, Ho VT, Bunin N, Iacobelli M, Liang W, Hume R, Tappe W, Soiffer R, Richardson P. Final results from a defibrotide treatment-IND study for patients with hepatic veno-occlusive disease/sinusoidal obstruction syndrome. Br J Haematol. 2018 Jun;181(6):816-827. doi: 10.1111/bjh.15267. Epub 2018 May 16. PMID 29767845

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Defibrotide
Started | 1206
Completed | 1154
Not Completed | 52

BASELINE CHARACTERISTICS:
Population: Safety Population
Arm/Group | Defibrotide
Number analyzed (Participants) | 1154
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at time of HSCT/chemo
  years | 19.32 (20.004)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 503
  Male | 651

OUTCOME MEASURES:

1. Primary Outcome: Survival by Day+100 Post Stem Cell Transplant or Chemotherapy
Time Frame: Day +100 from HSCT or 100 days from start of chemotherapy
Population: ITT Efficacy Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants alive
Arm/Group | Defibrotide
Number analyzed (Participants) | 571
Percentage of participants alive | 49.9 [45.8 to 54.0]

ADVERSE EVENTS:
Arm/Group | Defibrotide
Serious Adverse Events (participants affected / at risk) | 598/1154
Other Adverse Events (participants affected / at risk) | 166/1154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Defibrotide (N=1154)
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Coagulopathy (Blood and lymphatic system disorders) | 5
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Haemolysis (Blood and lymphatic system disorders) | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 13
Cardio-respiratory arrest (Cardiac disorders) | 9
Atrial flutter (Cardiac disorders) | 8
Pericardial effusion (Cardiac disorders) | 8
Bradycardia (Cardiac disorders) | 6
Atrial fibrillation (Cardiac disorders) | 5
Cardiac failure (Cardiac disorders) | 4
Cardiopulmonary failure (Cardiac disorders) | 3
Sinus bradycardia (Cardiac disorders) | 3
Cardiac tamponade (Cardiac disorders) | 2
Cardiomyopathy (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Atrial thrombosis (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 1
Torsade de pointes (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Retinal haemorrhage (Eye disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 33
Diarrhoea (Gastrointestinal disorders) | 9
Gastric haemorrhage (Gastrointestinal disorders) | 8
Ascites (Gastrointestinal disorders) | 7
Peritoneal haemorrhage (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 4
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 3
Mouth haemorrhage (Gastrointestinal disorders) | 3
Pneumatosis intestinalis (Gastrointestinal disorders) | 3
Rectal haemorrhage (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 2
Haematemesis (Gastrointestinal disorders) | 2
Abdominal compartment syndrome (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1
Malabsorption (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Multi-organ failure (General disorders) | 139
Pyrexia (General disorders) | 11
Disease progression (General disorders) | 2
Asthenia (General disorders) | 1
Catheter site haemorrhage (General disorders) | 1
Mucosal haemorrhage (General disorders) | 1
Multi-organ disorder (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pneumatosis (General disorders) | 1
Venoocclusive liver disease (Hepatobiliary disorders) | 87
Hepatic failure (Hepatobiliary disorders) | 19
Cholecystitis (Hepatobiliary disorders) | 4
Hepatorenal syndrome (Hepatobiliary disorders) | 3
Hepatic function abnormal (Hepatobiliary disorders) | 2
Acute hepatic failure (Hepatobiliary disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatorenal failure (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1
Graft versus host disease (Immune system disorders) | 15
Acute graft versus host disease (Immune system disorders) | 6
Graft versus host disease in intestine (Immune system disorders) | 6
Graft versus host disease in liver (Immune system disorders) | 5
Graft versus host disease in skin (Immune system disorders) | 3
Acute graft versus host disease in intestine (Immune system disorders) | 1
Acute graft versus host disease in liver (Immune system disorders) | 1
Acute graft versus host disease in skin (Immune system disorders) | 1
Engraftment syndrome (Immune system disorders) | 1
Sepsis (Injury, poisoning and procedural complications) | 32
Infection (Infections and infestations) | 17
Pneumonia (Infections and infestations) | 14
Septic shock (Infections and infestations) | 8
Lung infection (Infections and infestations) | 7
Cytomegalovirus infection (Infections and infestations) | 5
Bacteraemia (Infections and infestations) | 4
Pneumonia cytomegaloviral (Infections and infestations) | 4
BK virus infection (Infections and infestations) | 3
Bacterial sepsis (Infections and infestations) | 3
Device related infection (Infections and infestations) | 3
Pseudomonal bacteraemia (Infections and infestations) | 3
Sepsis syndrome (Infections and infestations) | 2
Staphylococcal bacteraemia (Infections and infestations) | 2
Staphylococcal infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Abdominal abscess (Infections and infestations) | 1
Abscess (Infections and infestations) | 1
Acid fast bacilli infection (Infections and infestations) | 1
Adenovirus infection (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Aspergillosis (Infections and infestations) | 1
Burkholderia cepacia complex infection (Infections and infestations) | 1
Candida sepsis (Infections and infestations) | 1
Cerebral fungal infection (Infections and infestations) | 1
Citrobacter sepsis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Corona virus infection (Infections and infestations) | 1
Enterobacter bacteraemia (Infections and infestations) | 1
Enterobacter infection (Infections and infestations) | 1
Enterococcal bacteraemia (Infections and infestations) | 1
Enterococcal infection (Infections and infestations) | 1
Enterococcal sepsis (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Fungal sepsis (Infections and infestations) | 1
Hepatitis viral (Infections and infestations) | 1
Human herpesvirus 6 infection (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Neutropenic infection (Infections and infestations) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1
Pneumonia parainfluenzae viral (Infections and infestations) | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 1
Pseudomonal sepsis (Infections and infestations) | 1
Pseudomonas infection (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Septic embolus (Infections and infestations) | 1
Stenotrophomonas sepsis (Infections and infestations) | 1
Systemic candida (Infections and infestations) | 1
Toxoplasmosis (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Zygomycosis (Infections and infestations) | 1
Transplant failure (Injury, poisoning and procedural complications) | 5
Procedural haemorrhage (Injury, poisoning and procedural complications) | 3
Brain herniation (Injury, poisoning and procedural complications) | 2
Engraft failure (Injury, poisoning and procedural complications) | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 2
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1
Feeding tube complication (Injury, poisoning and procedural complications) | 1
Hepatic haematoma (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1
Procedural complication (Injury, poisoning and procedural complications) | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 1
Urine output decreased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Transaminases increased (Investigations) | 2
Activated partial thromboplastin time prolonged (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Human herpes virus 6 serology positive (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Oxygen saturation decreased (Investigations) | 1
Pulse absent (Investigations) | 1
Weight increased (Investigations) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 6
Hypernatraemia (Metabolism and nutrition disorders) | 5
Acidosis (Metabolism and nutrition disorders) | 3
Fluid overload (Metabolism and nutrition disorders) | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hyperammonaemia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 2
Alkalosis (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Burkitt's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroblastoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Recurrent cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
T-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Encephalopathy (Nervous system disorders) | 9
Haemorrhage intracranial (Nervous system disorders) | 6
Convulsion (Nervous system disorders) | 5
Cerebral ischaemia (Nervous system disorders) | 3
Hepatic encephalopathy (Nervous system disorders) | 3
Hydrocephalus (Nervous system disorders) | 3
Subarachnoid haemorrhage (Nervous system disorders) | 3
Central nervous system haemorrhage (Nervous system disorders) | 2
Cerebral haemorrhage (Nervous system disorders) | 2
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 2
Autonomic neuropathy (Nervous system disorders) | 1
Brain hypoxia (Nervous system disorders) | 1
Brain injury (Nervous system disorders) | 1
Brain oedema (Nervous system disorders) | 1
Cerebellar haematoma (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
Hypertonia (Nervous system disorders) | 1
Intraventricular haemorrhage (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 45
Renal failure acute (Renal and urinary disorders) | 22
Cystitis haemorrhagic (Renal and urinary disorders) | 6
Renal impairment (Renal and urinary disorders) | 2
Azotaemia (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urogenital haemorrhage (Renal and urinary disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 80
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 57
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 31
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 22
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 16
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 6
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4
Apnoea (Respiratory, thoracic and mediastinal disorders) | 3
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2
Diffuse alveolar damage (Respiratory, thoracic and mediastinal disorders) | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2
Alveolar proteinosis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary veno-occlusive disease (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 46
Venoocclusive disease (Vascular disorders) | 9
Haemorrhage (Vascular disorders) | 7
Hypertension (Vascular disorders) | 4
Circulatory collapse (Vascular disorders) | 2
Haematoma (Vascular disorders) | 2
Hypovolaemic shock (Vascular disorders) | 2
Capillary leak syndrome (Vascular disorders) | 1
Catheter site haemorrhage (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
Haemorrhagic infarction (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Microangiopathy (Vascular disorders) | 1
Shock (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Defibrotide (N=1154)
Hypotension (Vascular disorders) | 93
Diarrhoea (Gastrointestinal disorders) | 70
Vomiting (Gastrointestinal disorders) | 63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No